CLINICAL TRIAL: NCT04761328
Title: Distress Associated With Stopping Immunotherapy of Cancer Patients
Brief Title: Fear of Recurrence and Stopping Immunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer Steel, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY19110214
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Behavioral Therapy
Keywords: Fear of recurrence; Quality of life; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: All patients will receive treatment and be evaluated pre- and post-treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cessation of treatment (Experimental): If the patient is randomized to this arm, they will be asked to stop their immunotherapy
  Interventions: Behavioral: cognitive behavioral therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — Cognitive-behavioral therapy involves changing these erroneous cognitions and beliefs through cognitive restructuring, modification of behavior, and development of alternative coping skills.

SUMMARY:
The study includes participants experiencing distress with regard to stopping immunotherapy and will utilize cognitive-behavioral therapy to reduce fear of recurrence, depression, and anxiety and improve quality of life.

DETAILED DESCRIPTION:
The intervention will be delivered through telemedicine to reduce the patient-related barriers to treatment including cost, transportation, and being able to maintain appointments while managing the side effects of treatment. The intervention will provide the patient with skills to reduce distress associated with ceasing treatment of a checkpoint inhibitor through the development evidence-based psychological and behavioral strategies that are tailored to the patients' preferences.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and older
* Fluent in English
* Diagnosis of cancer and history of treatment with immunotherapy

Exclusion Criteria:

* Active suicidal ideation, delusions or hallucinations

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduce fear of recurrence | 3 months
  Change by 50%

SECONDARY OUTCOMES:
Improve quality of life | 3 months
  Change of quality of life by 5 points
Reduction of anxiety | 3 months
  Change of anxiety by 2 points
Depressive symptoms | 3 months
  Change by 25%

CONTACTS AND LOCATIONS:
Overall Officials: Jason Luke, Principal Investigator — Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Centers, Pittsburgh, Pennsylvania, United States